CLINICAL TRIAL: NCT04563182
Title: Relationship Between Gluteus Medius Muscle Strength, Balance and Jumping Performance in Professional Female Handball Players
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Collaborators: Cyprus International University (Other)
Responsible Party: Principal Investigator, caglar soylu, Çağlar Soylu (Principal Investigator), Ankara Yildirim Beyazıt University
Other Study IDs: 2020-244
Record Dates: First submitted 2020-09-21; First posted 2020-09-24 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Gluteus Medius Muscle Strength; Handball Players; Balance; Jumping Performance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Muscle strength: GMed strength was assessed with the use of a Lafayette Manual Muscle Tester (Lafayette Instruments; Lafayette, Indiana, USA).
- Horizontal Jumping Performance: Lower extremity horizontal jumping was measured using the single leg hop (SLH) test as previously described
- Vertical Jumping Performance: To measure the single-leg vertical jump (SLVJ), the participants stood on the ground with their foot flat distributing their weight evenly on both feet.
- Dynamic Balance: The Y-Balance Test (YBT) was used to dynamic balance
- Static Balance: The Stork balance test (SBT) was used to measure static balance performance

SUMMARY:
Background Balance and jumping mechanisms are important to prevent injuries in sports such as handball, which require immediately change of direction, jumping and landing strategy. Strong proximal stability is required for accurate jump performance and stability.

Objective To investigate the relationship between gluteus medius strength and static, dynamic balance, horizontal and vertical jump performance.

Design Prospective field trial study.

Setting: Elite women handball players in Turkish Handball Super League. Patients (or Participants): Forty-two elite women handball players from Turkish Handball Super League were included in this study.

Interventions (or assessment of risk factors) The Lafayette Hand-Held Dynamometer was used to determine the strength of the gluteus medius. Single leg hop (SLH) test was used for horizontal jump and Lafayette Vertimetric device was used for vertical jump (VJ) evaluation. Y Balance Test (YBT) was used for the dynamic balance with direction of anterior, posteriomedial, posteriolateral and Standing Stork Test (SST) with eyes closed for the measurement of static balance.

Main outcome measurements Gluteus medius strength with hand dynamometer compared with YBT, SST, VJ and SLH tests.

ELIGIBILITY:
Inclusion Criteria:

* age between 18-40 years,
* playing Handball at least for 5 year as a professional player
* currently free of any lower limb injuries within the last three months
* no previous history of injury or surgery that may affect their lower limbs.

Exclusion Criteria:

* having lower limb injury for more than 1 month;
* having a history of surgery, or chronic and progressive disease in their lower limb
* having scoliosis or any other orthopaedic or neurological problems

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Thirty-nine professional female handball players from Turkish Handball Super League were included in this study
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-17 (Actual)

PRIMARY OUTCOMES:
Muscle strength | 2 weeks
  GMed strength was assessed with the use of a Lafayette Manual Muscle Tester (Lafayette Instruments; Lafayette, Indiana, USA).
Horizontal Jumping Performance | 2 weeks
  Lower extremity horizontal jumping was measured using the single leg hop (SLH) test as previously described
Vertical Jumping Performance | 2 weeks
  To measure the single-leg vertical jump (SLVJ), the participants stood on the ground with their foot flat distributing their weight evenly on both feet.
Dynamic Balance | 2 weeks
  The Y-Balance Test (YBT) was used to dynamic balance
Static Balance | 2 weeks
  The Stork balance test (SBT) was used to measure static balance performance

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Etlik, Turkey (Türkiye)